CLINICAL TRIAL: NCT06593938
Title: A Multicenter, Randomized, Open-label, Active-comparator Controlled Phase III Study to Evaluate the Efficacy and Safety of HRS-5965 Capsule in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Study to Evaluate the Efficacy and Safety of Oral HRS-5965 in Adult Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients Who Are Naive to Complement Inhibitor Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-301
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-5965 capsule (Experimental)
  Interventions: Drug: HRS-5965 capsule
- Eculizumab Injection (Experimental)
  Interventions: Drug: Eculizumab Injection

INTERVENTIONS:
Drug: HRS-5965 capsule — HRS-5965 capsule for 24 weeks
  Arms: HRS-5965 capsule
Drug: Eculizumab Injection — Eculizumab Injection for 24 weeks
  Arms: Eculizumab Injection

SUMMARY:
A study of the efficacy and safety of HRS-5965 capsules compared to eculizumab for 24 weeks in patients with PNH.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PNH confirmed by flow cytometry with clone size > 10%.
2. Have not received complement inhibitor therapy;
3. LDH > 1.5*ULN at screening.
4. Hemoglobin level < 10 g/dL at screening.

Exclusion Criteria:

1. Known or suspected hereditary or acquired complement deficiency;
2. Patients with laboratory evidence of bone marrow failure (reticulocytes <100x109/L; platelets <30x109/L; neutrophils <0.5x109/L);
3. Presence or suspicion of a systemic active bacterial, viral, or fungal infection (based on judgment of the investigator) within 2 weeks prior to the first dose of HRS-5965;
4. History of infection with capsular bacteria (e.g., meningococcus, pneumococcus, etc.)
5. Positive of HIV, HBsAg or HCVAb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with the hemoglobin levels are ≥ 12 g/dL at least on three out of four measurements in the absence of red blood cell transfusions | 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects with the change from baseline in hemoglobin is ≥ 2 g/dL at least on three out of four measurements in the absence of red blood cell transfusions | 24 weeks
Proportion of subjects who absence of administration of red blood cell transfusions | 24 weeks
Mean change from baseline in hemoglobin | 24 weeks
Mean percent change from baseline in LDH levels | 24 weeks
Mean change from baseline in reticulocyte counts | 24 weeks
Mean change from baseline in FACIT-Fatigue scores | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Blood Disease Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided